CLINICAL TRIAL: NCT01544842
Title: Comparison of Topical Tacrolimus, Triamcinolone and Placebo in the Treatment of Symptomatic Oral Lichen Planus
Brief Title: Tacrolimus Ointment in Oral Lichen Planus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources
Sponsor: University of Oulu (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Takrolimuusi123
Record Dates: First submitted 2012-01-04; First posted 2012-03-06 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2014-12

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; Tacrolimus ointment; Triamcinolone paste
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tacrolimus (Active Comparator): Tacrolimus ointment 0.1%, three times a day for 6-9 weeks.
  Interventions: Drug: 0.1 % tacrolimus ointment
- Triamcinolone (Active Comparator): Triamcinolone paste 0.1%, three times a day for 3-6 weeks.
  Interventions: Drug: 0.1 % triamcinolone paste
- Placebo (Placebo Comparator): Orabase paste, three times a day for 3-6 weeks.
  Interventions: Drug: Orabase paste

INTERVENTIONS:
Drug: 0.1 % tacrolimus ointment — applied topically to oral mucosa
  Other Names: Protopic
  Arms: Tacrolimus
Drug: 0.1 % triamcinolone paste — applied topically to oral mucosa
  Other Names: Kenacort-T paste, Kenacort-A paste
  Arms: Triamcinolone
Drug: Orabase paste — applied topically to oral mucosa
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of topical tacrolimus, triamcinolone and placebo in alleviating signs and symptoms of oral lichen planus (OLP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OLP made by a specialist in oral pathology based on clinical and histopathological features
* Clinical score for OLP ≥ 20 at baseline
* Symptomatic OLP at baseline
* Washout period of 2 weeks
* Age over 18

Exclusion Criteria:

* Pregnant or lactating women
* Allergy to tacrolimus or other macrolides
* Allergy to other drugs or substances used in the study
* Abnormal liver function
* Netherton's syndrome
* Cyclosporin medication
* Other regular medication that could have significant interactions with tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in clinical score for OLP | 1,2,3,4,5,6,7,8 and 9 weeks, 6 months
  The clinical score for OLP is a measure designed by the investigators for assessing the clinical extent and type of OLP, and the symptoms experienced by the patient. The value of the score is between 0-120.

CONTACTS AND LOCATIONS:
Overall Officials: Tuula Salo, DDS, PhD, Principal Investigator — Department of Diagnostics and Oral Medicine, Institute of Dentistry, University of Oulu, Oulu, Finland
Locations (2):
- Finland (2):
  - Oral and Maxillofacial Diseases Clinic, Kuopio University Hospital, Kuopio
  - Department of Diagnostics and Oral Medicine, Institute of Dentistry, University of Oulu, Oulu